CLINICAL TRIAL: NCT03900455
Title: Effectiveness of the Use of a Polyurethane Foam Multilayer Dressing in the Sacral Area, in Addition to Standard Healthcare, to Prevent the Onset of Pressure Ulcer in Patients at Risk. Multicentric Randomized Controlled Trial
Brief Title: Prevention of Pressure Ulcer on the Sacrum
Acronym: Multischiume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Multischiume
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Pressure Ulcer Risk
Keywords: Patients at risk; polyurethane foam; pressure ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocellular polyurethane foam multilayer dressing (Experimental)
  Interventions: Device: Hydrocellular polyurethane foam multilayer dressing; Procedure: Standard preventive care
- standard preventive care (Active Comparator)
  Interventions: Procedure: Standard preventive care

INTERVENTIONS:
Device: Hydrocellular polyurethane foam multilayer dressing — Application of a multilayer foam with 4 flaps that can be adapted to several areas of the body (including the sacrum) and consists of: an external polyurethane film, which is impermeable to liquids and bacteria using dynamic transpiration, which can form an impenetrable barrier to protect the skin; a protective layer that shields the skin against accidental knocks and helps to spread the pressure; a highly absorbent and leak-proof layer that traps the exudate inside; a layer of hydrocellular polyurethane foam; and, finally, in contact with the skin, a perforated evenly covered layer of silicone gel adhesive. in addition to Standard preventive care
  Other Names: ALLEVYN LIFE
  Arms: Hydrocellular polyurethane foam multilayer dressing
Procedure: Standard preventive care — Pressure Ulcer risk assessment using the Braden scale within 8 hours of admission. Place patient on pressure mattress (static or alternating pressure) if Braden score <17, daily inspection of the skin in the various pressure points and moving the patient at list every 4 hours. Management of possible incontinence, humidity control and prevention of skin damage and rubbing/friction during postural changes as per hospital procedure

SUMMARY:
The aim of the present study was to assess whether the application of a multilayered dressing made of hydrocellular polyurethane foam conformed to the sacral area (MSP) in addition to standard preventive care reduces the rate of pressure ulcer (PU) and their severity in population at risk admitted in acute care Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients at risk to develop Pressure Ulcer (Braden scale <17)
* without sacrum Pressure Ulcer
* Patients or legal guardians who give their consent to take part in the study

Exclusion Criteria:

* Patients with known allergy to the product being tested or dermatological diseases that prevent the use of topical products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Rate of any type of pressure ulcer in the sacral area. | On the seventh day of hospitalization or upon discharge from hospital, if that occurs before the seventh day
  The ulcer will be classified according to the National Pressure Ulcers Advisory Panel Classification. Pressure ulcer are classified and described through the use of staging systems. Staging systems describe the extent of tissue loss and the physical appearance of the injury caused by pressure and/or shear. From stage 1 (intact skin) to Stage 4 (Full-thickness skin and tissue loss).

SECONDARY OUTCOMES:
Pressure Ulcer Rate in the Sacral Area of Category≥ II | On the seventh day of hospitalization or upon discharge from hospital, if that occurs before the seventh day
  The ulcer will be classified according to the National Pressure Ulcers Advisory Panel Classification. Pressure ulcer are classified and described through the use of staging systems. Staging systems describe the extent of tissue loss and the physical appearance of the injury caused by pressure and/or shear. From stage 1 (intact skin) to Stage 4 (Full-thickness skin and tissue loss).
Skin irritation/damage due to the adhesive dressing | On the seventh day of hospitalization or upon discharge from hospital, if that occurs before the seventh day
  Clinical evaluation. It refers to any sort of inflammation and/or discoloration that distorts the skin's normal appearance. The skin may become scaly, bumpy, itchy, or otherwise irritated.
Number of dressing used per patient. | On the seventh day of hospitalization or upon discharge from hospital, if that occurs before the seventh day

CONTACTS AND LOCATIONS:
Locations (9):
- Italy (9):
  - ASO Azienda Ospedaliera Nazionale SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - Ausl Bologna Ospedale Maggiore, Bologna
  - Policlinico di S.Orsola Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - Ausl della Romagna, Cesena
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda USL- IRCCS di Reggio Emilia, Reggio Emilia
  - Policlinico Universitario Campus Bio-Medico di Roma, Roma
  - APSS Trento, Trento
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona

REFERENCES:
- [Derived] Forni C, Gazineo D, Allegrini E, Bolgeo T, Brugnolli A, Canzan F, Chiari P, Evangelista A, Grugnetti AM, Grugnetti G, Guberti M, Matarese M, Mezzalira E, Pierboni L, Prosperi L, Sofritti B, Tovazzi C, Vincenzi S, Zambiasi P, Zoffoli C, Ambrosi E; Multischiume Group. Effectiveness of a multi-layer silicone-adhesive polyurethane foam dressing as prevention for sacral pressure ulcers in at-risk in-patients: Randomized controlled trial. Int J Nurs Stud. 2022 Mar;127:104172. doi: 10.1016/j.ijnurstu.2022.104172. Epub 2022 Jan 8. PMID 35124474

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT03900455/Prot_SAP_ICF_000.pdf